CLINICAL TRIAL: NCT06727435
Title: Efficacy and Safety of Non-sedation Trial in Patients After Neurosurgical Craniotomy: a Single-arm, Single-centre Prospective Study
Brief Title: Efficacy and Safety of Non-sedation Trial in Patients After Neurosurgical Craniotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Guangzhi Shi, Director of the department of critical care unit, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: non-sedation trials
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Craniotomy; Neurosurgical Patients
Keywords: analgesia; sedation; craniotomy; neurosurgical patients
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: single-arm, single center, prospective clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- non-sedation strategy (Experimental): Patients eligible for this study will undergo non-sedation strategy, which continuous analgesia without sedation is performed with remifentanil. The remifentanil will be titrated (from 0.1µg/kg/min to 0.2ug/kg/min) every 10-15 minutes to achieve the goal for sedation (RASS score maintaining -2 to + 1). The patients in the non-sedation trial do not receive any sedatives but could receive bolus doses (2.5 or 5mg) of morphine for analgesia.
  Interventions: Drug: non-sedation strategy

INTERVENTIONS:
Drug: non-sedation strategy — Patients eligible for this study will undergo non-sedation strategy, which continuous analgesia without sedation is performed with remifentanil. The remifentanil will be titrated (from 0.1µg/kg/min to 0.2ug/kg/min) every 10-15 minutes to achieve the goal for sedation (RASS score maintaining -2 to + 1). The patients in the non-sedation trial do not receive any sedatives but could receive bolus doses (2.5 or 5mg) of morphine for analgesia.

SUMMARY:
Neurosurgical patients may be more vulnerable to stress caused by agitation after craniotomy, due to longer anesthesia duration, delayed extubation and pain and post-craniotomy frontal pneumocephalus and so on. Analgesia and sedation are important to the neurosurgical patients. However, there is little data to document the effects of protocolised analgesia and sedation on patients with neurological injury. The analgesia and sedation for neurosurgical patients is complex and difficult. The aim of the study is to explore the efficacy and safety of non-sedation strategies in patients admitted to ICU after neurosurgery craniotomy. This is a single-arm, single center, prospective clinical trial. Sixty- five adult patients whose Richmond Agitation-Sedation Scale (RASS) score greater than 1 point and intensive care unit (ICU) stay > 24 hours after neurosurgical craniotomy will be enrolled. Patients eligible for this study will undergo non-sedation strategy, which continuous analgesia without sedation is performed with remifentanil. The remifentanil will be titrated (from 0.1µg/kg/min to 0.2ug/kg/min) every 10-15 minutes to achieve the goal for sedation (RASS score maintaining -2 to + 1). The patients in the non-sedation trial do not receive any sedatives but could receive bolus doses (2.5 or 5mg) of morphine for analgesia. The primary endpoints is the rate of successful sedation using non-sedation trials in the patients after neurosurgical craniotomy in ICU, defined as 1) RASS score -2 to +1. 2) No additional sedation required (any sedation medicine). The safety endpoints are the incidence of adverse events, including accidental removal of tubes (tracheal reintubation within 2 hours after extubation and reintubation of central venous catheterization (CVC) or gastric tube within 4h), significant agitation (RSAA score greater than 2), occurrences of need for CT or MRI brain scans.

DETAILED DESCRIPTION:
In the intensive care unit (ICU), analgesia and sedation treatment is an important part of the clinical management for patients. The aim of the analgesia and sedation includes reducing pain of the disease or catheters, controlling anxiety, reducing stress response, improving the coordination of mechanical ventilation, and reducing the noxious stimulation . After craniotomy, the patients always are admitted to ICU. And postoperative agitation after general anesthesia may be associated with serious consequences, such as unplanned extubation, injuries and longer post-anesthesia care unit stay. The incidence of agitation after elective intracranial operations was 29%, which was higher than that previously observed in other surgical populations. Neurosurgical patients may be more vulnerable to stress caused by agitation, due to longer anesthesia duration, delayed extubation and pain and post-craniotomy frontal pneumocephalus. Brain lesions and intracranial manipulations in neurosurgical patients might affect the brain regions which involves cognition and emotion, and are assumed to influence postoperative cognition.

However, the investigations of analgesia and sedation in neurosurgical populations have been inadequate. Most of the researches about analgesia and sedation in ICU were excluded the neurosurgical patients. These patients are special for its cruciality of evaluating the consciousness and neurological signs examination. The analgesia and sedation management is difficult. Recent years, a single-center study showed that non-sedation group had more days without mechanical ventilation and shorter stay in ICU. Non-sedation provides a new way for analgesia and sedation. Moreover, during our clinical work, we noticed that non-sedation trial may serve as a useful project to remit agitation in patients after neurosurgical craniotomy. Considering the efficacy and safety of non-sedation trial in patients after neurosurgical craniotomy, further investigation is needed. Therefore, we conducted this single-arm, single-centre prospective study in the adult patients admitted to ICU after neurosurgery craniotomy. The aim of the study is to explore the efficacy and safety of non-sedation strategies in patients admitted to ICU after neurosurgery craniotomy, hoping to provide a new direction for analgesia and sedation of patients after neurosurgical craniotomy.

Study design This single-centre, single-arm, open-label clinical study will be conducted in the Department of Critical Care Unit, Beijng Tiantan Hospital, Capital Medical University in China, which is with a neurosurgery unit. ICU receives mainly neurocritical care patients after neurosurgical craniotomy. Meeting the screening criteria, the patients will be recruited to the study. The study is to explore the efficacy and safety of non-sedation trial in patients after neurosurgical craniotomy. This trial is reported according to the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) reporting guidelines.

Informed consent All the patients admitted in ICU after neurosurgical craniotomy will be screened. For inclusion, all patients will first need to provide written informed consent and orally receive detailed protocol instructions. Informed consent will include the purpose of the study, the necessary of analgesic and sedation, the advantages and disadvantages of the protocol, a list of possible adverse effects or risks associated with the treatment. Participants will also be informed that they could withdraw from the study at any time for any reason. No patient will participate in the study without the formal procedure of informed consent.

Inclusion criteria

1. Age: 18-85 years old, with ICU stay > 24 hours;
2. The Richmond Agitation-Sedation Scale (RASS) score is greater than 1 point (Restless: anxious or apprehensive but movements not aggressive or vigorous);
3. Patients after neurosurgical craniotomy. Exclusion criteria

1.Patients who need deep sedation (PaO2/FiO2≤100 mmHg, loss of consciousness during muscle relaxant therapy, status epilepticus, absolute braking for surgical or surgical conditions, severe traumatic brain injury and cranial hypertension, therapeutic hypothermia and other clinical assessments need to maintain RASS <-2); 2.Patients who may damage the medullary bullongans which contents respiratory center and avoid the application of analgesic drugs; 3.Patients who cannot assess the RASS score due to various reasons, such as aphasia, history of mental system (schizophrenia, mania, confusion, history of cognitive dysfunction), generalized seizure status, coma patients, postoperative aphasia, etc.; 4.Patients who use sedatives or opioid analgesics ≥ 1 week before enrollment; 5.The expected ICU stay time less than 24 hours; 6.The patients with delirium, alcohol withdrawal symptoms or mental illness or the use of antipsychotic drugs; 7.Severe abnormal liver function (Child-Pugh grade C); 8.Renal insufficiency requiring renal replacement therapy; 9.Surgical treatment is required during the ICU (except for short surgery, such as lumbar puncture, ventricular drainage, etc.); 10.Study drug allergy or other contraindications; 11.women during pregnancy or lactation; 12. Who was selected in other RCT tests; 13.The patient himself or the legally authorized person is not willing to participate in the trial; 14.The investigator judged that the patient is not suitable for inclusion (such as severe hypotension; potential disputes, etc.).

Study intervention All the patients admitted to ICU after neurosurgical craniotomy will be screened daily. The patient meeting the inclusion criteria will be included in the study. In the centre, the depth of sedation and pain will be routinely assessed by Richmond Agitation-Sedation Scale (RASS) and Critical Care Pain Observation Tool (CPOT), with targeted values of -2 to +1 and 0-1, respectively.

If the patients are uncomfortable, a doctor is consulted, and any possible causes for patient discomfort are investigated (eg, hypoxia, tube obstruction, pain). If needed, a person is assigned to verbally comfort and reassure the patient. Physical restraints were never used. If patients still feel uncomfortable with RASS score greater that 1 points, they will receive non-sedation trial.

Continuous analgesia without sedation is performed with remifentanil during the non-sedation trial. The initial dose of remifentanil is 6-9 µg/kg/h (0.1 to 0.15µg/kg/min), and the dose of remifentanil will be adjusted every 10-15min (1.025 ug/kg/min) to achieve optimal level of sedation. The maximal dose of remifentanil reaches 12 ug/kg/h (0.2ug/kg/min), excess remifentanil is not allowed[16]. The patients in the non-sedation trial do not receive any sedatives but could receive bolus doses (2.5 or 5mg) of morphine for analgesia. If the infusion rate is greater than 12 ug/kg/h(0.2ug/kg/min) and the infusion fails to meet the standard after intermittent analgesia administration, the patients are sedation with midazolam or propofol for safety and meeting the clinical needs. And if the clinician thinks sedation is necessary to ensure adequate oxygenation or placement in the prone position, the patient will be treated with the conventional analgesic sedation group. The goal for sedation was the RASS score of-2 to + 1.

Meanwhile, the delusion (CAM-ICU score) was assessed at 7:00 and 21:00 daily, and if treatment is required, the initial choice was to use non-pharmacological intervention (reassurance or mobilization). If not, medication is required, which may include haloperidol (1,2.5 or 5mg) or olanzapine.

Study medication: Rmifentanil hydrochloride for injection(Jiangsu Enhua Pharmaceutical Co., LTD., trade name Rufen), specification: 2mg, H20143315, Chinese drug approval, validity period of 24 months, 2-25℃.

Sample size In this study, the non-inferiority sample size calculation of Power Analysis and Sample Size (PASS) 15.0 software is used. The study is a non-inferiority, a single group design. And the primary endpoint is the rate of successful sedation using non-sedation trials in the patients after neurosurgical craniotomy in ICU. However, there is no reported data on the successful rate of non-sedation trial, we use the successful rate on conventional analgesia and sedation management, which is 99% as expected. Suppose the non-inferiority threshold is 5%, I error is 0.025 and the power of test is 80%. The required number of eligible samples is 61. Considering the drop rate of 5%, the study is expected to enrol 65 patients after neurosurgical craniotomy in ICU.

Statistical analysis In this study, the target population for the analysis is defined as a full analysis set (FAS). FAS is defined as the population of all enrolled patients excluding cases that will not meet the eligibility criteria. Patient characteristic data will be expressed as median (range). For items observed as discrete values, the number of examples in each category and their proportions will be calculated using summary statistics. Time-to-event data, including cost in ICU, the duration of intubation, days without mechanical ventilation, length of stay in the ICU, length of hospital stay, mortality in hospital, will be calculated using the Kaplan-Meier method. Statistical tests for the main analysis will be performed at a two-tailed 5% significance level. Statistical significance is defined by a p value<0.05. All analyses will be performed using IBM SPSS (SPSS,24.0) software.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-85 years old, with ICU stay > 24 hours;
* The Richmond Agitation-Sedation Scale (RASS) score is greater than 1 point (Restless: anxious or apprehensive but movements not aggressive or vigorous);
* Patients after neurosurgical craniotomy.

Exclusion Criteria:

* Patients who need deep sedation (PaO2/FiO2≤100 mmHg, loss of consciousness during muscle relaxant therapy, status epilepticus, absolute braking for surgical or surgical conditions, severe traumatic brain injury and cranial hypertension, therapeutic hypothermia and other clinical assessments need to maintain RASS <-2);
* Patients who may damage the medullary bullongans which contents respiratory center and avoid the application of analgesic drugs;
* Patients who cannot assess the RASS score due to various reasons, such as aphasia, history of mental system (schizophrenia, mania, confusion, history of cognitive dysfunction), generalized seizure status, coma patients, postoperative aphasia, etc.;
* Patients who use sedatives or opioid analgesics ≥ 1 week before enrollment;
* The expected ICU stay time less than 24 hours;
* The patients with delirium, alcohol withdrawal symptoms or mental illness or the use of antipsychotic drugs;
* Severe abnormal liver function (Child-Pugh grade C);
* Renal insufficiency requiring renal replacement therapy;
* Surgical treatment is required during the ICU (except for short surgery, such as lumbar puncture, ventricular drainage, etc.);
* Study drug allergy or other contraindications;
* women during pregnancy or lactation;
* Who was selected in other RCT tests;
* The patient himself or the legally authorized person is not willing to participate in the trial;
* The investigator judged that the patient is not suitable for inclusion (such as severe hypotension; potential disputes, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoints is the efficacy and safety of non-sedation trial | from enrollment to the discharge of ICU, 28 days or death, whichever came first
  The primary endpoints is the rate of successful sedation using non-sedation trials in the patients after neurosurgical craniotomy in ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, South 4th Ring West Road 119, Fengtai District, Beijing 100070, China., Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used in this study will be available from the corresponding author on reasonable request.